CLINICAL TRIAL: NCT01803139
Title: Long Term Outcomes of a Multicentre Controlled Clinical Trial of Breast Irradiation Using Intensity-Modulated Radiation Therapy
Brief Title: Long Term Results of the Canadian Breast IMRT Study
Acronym: IMRT-FU
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMRT-02
Record Dates: First submitted 2012-03-01; First posted 2013-03-04 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Breast Cancer
Keywords: Breast cancer radiotherapy IMRT
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard breast radiotherapy (Active Comparator): The treatment is planned using 2D wedges optimisation on the central CT-planning slice.
  Interventions: Device: Adjuvant breast radiotherapy
- Breast IMRT (Experimental): The treatment is planned 3D IMRT optimisation using all CT-planning slices.
  Interventions: Device: Adjuvant breast radiotherapy

INTERVENTIONS:
Device: Adjuvant breast radiotherapy — Adjuvant radiotherapy delivering 50 Gy in 25 treatments, with an additional boost dose of 16 Gy at the discretion of the radiation oncologist.
  Other Names: Intensity Modulated Radiation Therapy

SUMMARY:
Women diagnosed with an early stage cancer of the breast usually have the cancer removed by lumpectomy and then have radiation treatments to the entire breast. In 2008 the investigators published the result of a multicentre study showing that breast Intensity Modulated Radiation Therapy (IMRT) significantly reduces the occurrence of radiation burns. In this study the investigators will recall all patients at 8 years to assess if this technique also reduces permanent side effects including pain and cosmesis.

DETAILED DESCRIPTION:
In 2008 our group published the results of a multicentre, randomized, double-blinded study comparing standard radiotherapy to breast IMRT. The study showed a significant reduction moist desquamation using breast IMRT from 47.8% to 31.2% (p=0.002). There are two other Phase III trials showing improvement of long term cosmetic outcomes. Yet the use of breast IMRT remains not widely accepted. This trial aims at evaluating long term tolerance of breast IMRT compared to standard radiotherapy.

The investigators hypothesize that breast IMRT reduces the occurence of chronic breast pain (primary objective), improves cosmesis, reduces the occurence of delayed and permanent radiation induced skin side effects (telangiectasia, dryness, induration, edema, discolorations), improves quality of life. The investigators also hypothesize that there will not be differences in the local control rate or survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated in the Canadian Phase 3 randomised controlled trial breast IMRT trial

Exclusion Criteria:

* Patients declining participating to this study
* Patients unable to travel to the study site
* Patients deceased

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Chronic breast pain using Visual Analog Scale | 8 years plus or minus one year
  Quantitatively patients will be asked if they have spontaneous breast pain in the treated breast during the last 6 months, and will be asked to rate its intensity using a Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (extreme pain).
Chronic breast pain using the Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE 4.0) | 8 years plus or minus one year
  Quantitatively pain intensity will be evaluated using the Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE 4.0).
Chronic breast pain using the prescription of pain killer | 8 years plus or minus one year
  The use of pain killer will be recorded.
Chronic breast pain using the McGill pain questionnaire | 8 years plus or minus one year
  Qualitatively the pain will be evaluated and scored using the short form of the McGill pain questionnaire.

SECONDARY OUTCOMES:
Skin and sub-cutaneous delayed side effects using the European Organization for Research and Treatment of Cancer (EORTC) scale | 8 years plus or minus one year
  Skin and subcutaneous late radiation toxicity will be assessed by the clinical trial assistant using the European Organization for Research and Treatment of Cancer (EORTC) breast cancer rating system for the cosmesis assessment. This scale evaluates skin discoloration and oedema comparing between breasts as no, small, moderate or large differences.
Cosmesis using the Breast Cancer Treatment Outcome Scale (BCTOS) | 8 years plus or minus one year
  The patient's cosmesis self-report will be used as most reliable cosmetic endpoint and will use the Breast Cancer Treatment Outcome Scale (BCTOS).
Quality of Life using the European Organization for Research and Treatment of Cancer (EORTC) general module questionnaire (C-30) | 8 years plus or minus one year
  At time of initial treatment patient's quality of life was assessed at baseline, the last week of treatment, and 6 weeks after treatment using the European Organization for Research and Treatment of Cancer (EORTC) quality of life general module (C-30) self-assessment questionnaire. The same questionnaire will be administered to ensure consistency in the quality of life assessment and enable comparisons over time for individuals and cohorts.
Skin and sub-cutaneous delayed telangiectasia | 8 years plus or minus one year
  Telangiectasia will be classified into four categories of surface: none, less than 1cm2, 1 to 4 cm2 and over 4cm2.
Skin and sub-cutaneous induration | 8 years plus or minus one year
  Induration will be evaluated using the Late Radiation Morbidity Scoring Scheme scale that classifies fibrosis in four grades.
Cosmesis using the European Organization for Research and Treatment of Cancer (EORTC) scale | 8 years plus or minus one year
  Research assistant will use the four point scale European Organization for Research and Treatment of Cancer (EORTC) to evaluate cosmesis.
Cosmesis using digital photographs | 8 years plus or minus one year
  Digital photographs will be taken of the treated and untreated breasts and will be evaluated for cosmetic results by four blinded individuals using the EORTC criteria and the consensus score will be recorded.
Quality of Life using the European Organization for Research and Treatment of Cancer (EORTC) breast module questionnaire (BR-23) | 8 years plus or minus one year
  At time of initial treatment patient's quality of life was assessed at baseline, the last week of treatment, and 6 weeks after treatment using the European Organization for Research and Treatment of Cancer (EORTC) quality of life breast module (BR-23) self-assessment questionnaire. The same questionnaire will be administered to ensure consistency in the quality of life assessment and enable comparisons over time for individuals and cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Pignol, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - Vancouver Island Cancer Centre, Victoria, British Columbia
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario

REFERENCES:
- [Result] Pignol JP, Olivotto I, Rakovitch E, Gardner S, Sixel K, Beckham W, Vu TT, Truong P, Ackerman I, Paszat L. A multicenter randomized trial of breast intensity-modulated radiation therapy to reduce acute radiation dermatitis. J Clin Oncol. 2008 May 1;26(13):2085-92. doi: 10.1200/JCO.2007.15.2488. Epub 2008 Feb 19. PMID 18285602